CLINICAL TRIAL: NCT05922189
Title: The Effect of SBS Decompression Technique on Gastrointestinal Symptoms During Menstrual Cycle: a Single-blind Randomized Controlled Trial
Brief Title: The Effect of the SBS Decompression Technique on Gastrointestinal Symptoms During the Menstrual Cycle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OST1-006
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Gastrointestinal symptoms; Menstrual cycle; SBS decompression; Osteopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBS Decompression Technique (Experimental): The technique was preformed until the investigator felt a relaxation of the structures, with a maximum duration of 5 minutes.
  Interventions: Other: SBS Decompression Technique
- Placebo Technique (Placebo Comparator): The technique was preformed during 2 minutes.
  Interventions: Other: Placebo Technique

INTERVENTIONS:
Other: SBS Decompression Technique — The investigator who applied the technique stood on the right side, laterally to the headboard of the table, with feet flat on the floor, at an appropriate level in relation to the volunteer's headboard, and with a glove on his right hand. Then, he contacted the volunteer's sphenoid wings with his left hand and asked the volunteer to open her mouth, contacting the upper dental arch with the second and third fingers of his right hand. Subsequently, the investigator brought both hands together, followed by an inspiration towards the floor and then a translation towards the ceiling until he felt the structures relax, with a maximum duration of 5 minutes. A second Investigator was sitting on a chair, placed on the opposite side of the head of the table with a stopwatch in his dominant hand, in order to time the application time of each technique.
  Arms: SBS Decompression Technique
Other: Placebo Technique — The investigator was standing, on the right side, laterally to the headboard of the table with feet flat on the floor, at an appropriate level in relation to the headboard of the volunteer's and with a glove on his right hand. Then, he contacted the participant's sphenoid wings with his left hand and asked her to open her mouth. With the second and third fingers of the right hand, he made contact with the upper dental arch. These contacts were maintained for 2 minutes, without moving. A second investigator sat on a chair, placed on the opposite side of the table with the stopwatch in his dominant hand, in order to time the application time of each technique.
  Arms: Placebo Technique

SUMMARY:
Determining the effects of a single application of the sphenobasilar synchondrosis (SBS) decompression technique, on gastrointestinal symptoms during the menstrual cycle is an area that lacks of evidence and proper studies. Therefore the investigators consider this an interesting topic to study.

DETAILED DESCRIPTION:
The menstrual cycle is determined by cyclic changes in hormones levels, whose secretion is regulated by the feedback system of the hypothalamic-pituitary-gonadal axis and lasts approximately 28 days. These hormones have direct effects on organs as well as on the peripheral and central nervous systems (CNS), acting alone or in combination to influence both bowel function and gastrointestinal symptoms.

Premenstrually, uterine prostaglandin production can mediate an inflammatory response characterized by pain, and during menstruation, abnormally high levels of prostaglandins in menstrual fluid can induce abnormal uterine contractions. In the intestine, prostaglandins can cause smooth muscle contractions, as well as reduced absorption and induced secretion of electrolytes in the small intestine, increasing gastrointestinal symptomatology.

A study concluded that sphenobasilar synchondrosis (SBS) dysfunctions may be directly related to changes in the endocrine and hormonal system, due to the location of the pituitary gland (endocrine gland responsible for the release mainly of follicle stimulating hormone (FSH) and lutein hormone (LH)). Thus, there is a relationship between the SBS decompression technique and gastrointestinal symptoms during the menstrual cycle.

However this theme lacks of scientific evidence, therefore the investigators intend to collaborate to increase knowledge in this area, determining the effects of the SBS decompression technique, on gastrointestinal symptoms during the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Ages between 18 and 25 years old;
* Gastrointestinal symptoms in the week before, during, or after menstrual period;
* Regular menstrual cycle ;
* Taking an oral hormonal pill.

Exclusion Criteria:

* People who are undergoing / who have already undergone hormonal therapies;
* Pregnancy;
* Orthodontic braces or dental plate;
* Temporomandibular joint dysfunction or other dysfunction that prevents the opening of the mouth;
* Present or have presented in the last 3 months any of these conditions: high blood pressure, tumors, acute intracranial bleeding/haemorrhage, increased intracranial pressure, acute skull fracture, convulsive states;
* Started/changed/stopped taking a hormonal contraceptive method in the last 3 months;
* BMI greater than 30;
* Students of osteopathy or being subjected to an osteopathic treatment during the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in abdominal pain pre and post intervention | Two months after first intervention
  The participants were submited to constant evaluation through the diary that they had to fill in daily, during two menstrual cycles, which corresponds to a total of about 2 months. At the end of completing each cycle, the corresponding diary was sent to the researchers, so that they could record the information.
Change from baseline in number of bowel movements (per day) pre and post intervention | Two months after first intervention
  The participants were submited to constant evaluation through the diary that they had to fill in daily, during two menstrual cycles, which corresponds to a total of about 2 months. At the end of completing each cycle, the corresponding diary was sent to the researchers, so that they could record the information.
Change from baseline in type of feces pre and post intervention | Two months after first intervention
  The participants were submited to constant evaluation through the diary that they had to fill in daily, during two menstrual cycles, which corresponds to a total of about 2 months. At the end of completing each cycle, the corresponding diary was sent to the researchers, so that they could record the information.
Change from baseline in nausea pre and post intervention | Two months after first intervention
  The participants were submited to constant evaluation through the diary that they had to fill in daily, during two menstrual cycles, which corresponds to a total of about 2 months. At the end of completing each cycle, the corresponding diary was sent to the researchers, so that they could record the information.
Change from baseline in presence of abdominal distention pre and post intervention | Two months after first intervention
  The participants were submited to constant evaluation through the diary that they had to fill in daily, during two menstrual cycles, which corresponds to a total of about 2 months. At the end of completing each cycle, the corresponding diary was sent to the researchers, so that they could record the information.
Change from baseline in need to take laxatives pre and post intervention | Two months after first intervention
  The participants were submited to constant evaluation through the diary that they had to fill in daily, during two menstrual cycles, which corresponds to a total of about 2 months. At the end of completing each cycle, the corresponding diary was sent to the researchers, so that they could record the information.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Politécnico do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bharadwaj S, Kulkarni G, Shen B. Menstrual cycle, sex hormones in female inflammatory bowel disease patients with and without surgery. J Dig Dis. 2015 May;16(5):245-55. doi: 10.1111/1751-2980.12247. PMID 25851437
- [Background] Chang L, Heitkemper MM. Gender differences in irritable bowel syndrome. Gastroenterology. 2002 Nov;123(5):1686-701. doi: 10.1053/gast.2002.36603. PMID 12404243
- [Background] Dajani EZ, Shahwan TG, Dajani NE. Prostaglandins and brain-gut axis. J Physiol Pharmacol. 2003 Dec;54 Suppl 4:155-64. PMID 15075457
- [Background] Lim SM, Nam CM, Kim YN, Lee SA, Kim EH, Hong SP, Kim TI, Kim WH, Cheon JH. The effect of the menstrual cycle on inflammatory bowel disease: a prospective study. Gut Liver. 2013 Jan;7(1):51-7. doi: 10.5009/gnl.2013.7.1.51. Epub 2013 Jan 11. PMID 23423645
- [Background] Bernstein MT, Graff LA, Targownik LE, Downing K, Shafer LA, Rawsthorne P, Bernstein CN, Avery L. Gastrointestinal symptoms before and during menses in women with IBD. Aliment Pharmacol Ther. 2012 Jul;36(2):135-44. doi: 10.1111/j.1365-2036.2012.05155.x. Epub 2012 May 24. PMID 22621660
- [Background] Parlak E, Dagli U, Alkim C, Disibeyaz S, Tunc B, Ulker A, Sahin B. Pattern of gastrointestinal and psychosomatic symptoms across the menstrual cycle in women with inflammatory bowel disease. Turk J Gastroenterol. 2003 Dec;14(4):250-6. PMID 15048600
- [Background] Elhadd TA, Neary R, Abdu TA, Kennedy G, Hill A, McLaren M, Akber M, Belch JJ, Clayton RN. Influence of the hormonal changes during the normal menstrual cycle in healthy young women on soluble adhesion molecules, plasma homocysteine, free radical markers and lipoprotein fractions. Int Angiol. 2003 Sep;22(3):222-8. PMID 14612848